CLINICAL TRIAL: NCT00494546
Title: High Versus Low Dose Supplemental External Radiation With Pd-103 for Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: Schiffler Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2044
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2007-06

CONDITIONS: Prostate Cancer
Keywords: prostate; brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pd-103 with 20 vs 44 Gy supplemental beam XRT

SUMMARY:
Objective: The objective of this study is test the hypothesis that delivering a higher percentage of the radiation dose as external radiation versus implant will lead to higher tumor control rates.

Research design A total of 600 patients with AJC clinical stage T1-T2 prostatic carcinoma (Gleason grade 7 to 10 and/or PSA 10 to 20 ng/ml) will be randomized to treatment with 44 Gy versus 20 Gy external radiation plus a Pd-103 implant boost (90 Gy versus 105 Gy, respectively).

DETAILED DESCRIPTION:
Objective: The objective of this study is test the hypothesis that delivering a higher percentage of the radiation dose as external radiation versus implant will lead to higher tumor control rates.

Research design A total of 600 patients with AJC clinical stage T1-T2 prostatic carcinoma (Gleason grade 7 to 10 and/or PSA 10 to 20 ng/ml) will be randomized to treatment with 44 Gy versus 20 Gy external radiation plus a Pd-103 implant boost (90 Gy versus 105 Gy, respectively).

Methodology: Patients will be randomized by the method of random permuted blocks.

Cancer status will be monitored by serial serum PSA at 6, 12, 18 and 24 months and yearly thereafter. Treatment-related morbidity will be monitored by personal interview, using standard American Urologic Association and Radiation Therapy Oncology Group criteria at 1, 3, 6, 12 and 24 months. The primary endpoint will be based on serum PSA. A value above 1.0 ng/ml two years after treatment will be considered to have residual or recurrent cancer and to have failed therapy.

Findings: 566 patients have been randomized and the study was closed due to slowing accrual. A preliminary analysis shows similar morbidity between the treatment arms, and nearly identical cancer control rates between randomization arms.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Prostate cancer
* PSA 10-20
* Gleason score 7-10

Exclusion Criteria:

* Lymph nodes positive

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 1999-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
cancer control | 5-year post treatment

SECONDARY OUTCOMES:
rectal and urinary morbidity | 2- and 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Kent E Wallner, MD, Study Chair — Puget Sound Health Care system
Locations (1):
- VA Puget Sound, Seattle, Washington, United States

REFERENCES:
- [Result] Wallner K, Merrick G, True L, Sherertz T, Sutlief S, Cavanagh W, Butler W. 20 Gy versus 44 Gy supplemental beam radiation with Pd-103 prostate brachytherapy: preliminary biochemical outcomes from a prospective randomized multi-center trial. Radiother Oncol. 2005 Jun;75(3):307-10. doi: 10.1016/j.radonc.2005.03.019. PMID 16086912